CLINICAL TRIAL: NCT05363371
Title: A Mindfulness and Peer Mentoring Program to Improve Adherence to Medication Assisted Treatment for Opioid Use Disorders (R33 Phase)
Brief Title: Minds and Mentors Program- R33
Acronym: MiMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other); Tuscaloosa Veterans Affairs Medical Center (U.S. Federal Agency); Pathway Healthcare, LLC (Unknown)
Responsible Party: Principal Investigator, Mercy N. Mumba, Associate Professor of Nursing, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4R33AT010802-02 (NIH)
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Opioid Use Disorder; Substance Use Disorders; Medication Assisted Treatment
Keywords: Opioid Use Disorder; Mindfulness based therapy; Cravings; Relapse prevention; Treatment retention; Depression; Stress; Anxiety; Cortisol; Peer Mentors
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness based relapse prevention and peer mentoring (Experimental): Treatment will utilize a group format. The twelve-week mindfulness based relapsed prevention group therapy intervention is co-led by a licensed counselor and a peer mentor for eight weeks, followed by group sessions led by peer mentors for an additional four weeks.
  Interventions: Behavioral: Minds and Mentors
- 12 Step Treatment Program (Active Comparator): Participants in the attentional control group will attend 12 weeks of a enhanced 12 step treatment program.
  Interventions: Behavioral: Twelve Step Intervention Group

INTERVENTIONS:
Behavioral: Minds and Mentors — Participants will be randomized into Minds and Mentors to attend weekly group therapy sessions for 12 week. The mindfulness-based relapse prevention therapy intervention will be led by a licensed counselor for eights weeks followed up by four additional sessions led by a certified recovery support specialist (peer mentor).
  Arms: Mindfulness based relapse prevention and peer mentoring
Behavioral: Twelve Step Intervention Group — Participants will be randomized to the Twelve Step Intervention Group to attend weekly group therapy sessions for 12 week. The twelve step intervention group will be led by a licensed counselor.
  Arms: 12 Step Treatment Program

SUMMARY:
The proposed research effort will:

The purpose of this study is as follows:

1. Test the effectiveness of the Minds and Mentors Program in a group treatment trial in which individuals using medications for opioid use disorder (MOUD) will be randomized in blocks of five to receive either the Minds and Mentors Program (n=120) or Twelve Step Facilitation (n=120).
2. Determine whether the MiMP: a) improves adherence to MOUD b) reduces the rate of relapse and cravings c) decreases self-reported anxiety, stress, and depression and d) reduces cortisol levels and cortisol reactivity to drug cues.
3. Examine whether pre-intervention cortisol reactivity is predictive of relapse outcomes, and/ or reductions in cortisol reactivity over the course of intervention mediate relapse outcomes.

DETAILED DESCRIPTION:
Although medications for opioid use disorders (MOUD) is safe and effective and is currently considered the gold standard for treating OUD, adherence to MOUD regimens remains a challenge. Early studies have demonstrated efficacy of mindfulness-based interventions as adjunctive treatment for substance use disorders (SUD) while reducing substance use and cravings. In addition, non-randomized pilot studies suggest that mindfulness-based interventions may be effective in reducing symptoms of depression and anxiety in individuals undergoing MOUD.

The goal of the proposed study is to determine the effectiveness of a mindfulness-based intervention that also utilizes peer mentors in addition to professional substance abuse therapists (the Minds and Mentors program [MiMP]) in improving adherence to MOUD and reducing relapse rates in a sample of individuals with OUD who are also on MOUD versus a twelve-step facilitation (TSF) program. The MiMP is a twelve-week intervention that uses group therapy and meets once a week for about two hours. The primary outcome measure will is adherence to medications for OUD. The secondary outcome measures will include the demographic covariates, depression, anxiety, stress, quality of life, and cravings. Finally, exploratory outcome measures will include cortisol levels and rates of reactivity to drug cues. This study will randomize participants in either intervention or control group in blocks of five. Data collection will occur at baseline, 8 weeks, 12 weeks (end of treatment) and at 12- week and 24- week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 and older
2. Opioid Use disorder diagnosis based on DSM-V criteria in the past 30 days
3. Currently receiving MOUD (e.g. methadone, naloxone, naltrexone, and buprenorphine) from an established provider
4. Are within maintenance phase of MOUD (not actively detoxing)
5. May meet criteria for a mood, anxiety, or other psychiatric disorder based on the DSM-V criteria. Participants on maintenance medications for a mood or anxiety disorder must be stabilized on medications for at least 2 weeks before therapy initiation
6. Capable of reading and understanding English
7. Able to provide written informed consent (i.e. no surrogate)
8. Access to a smartphone or a computer with an internet connection
9. Willing to commit to 12 group therapy sessions, baseline, and follow-up assessments for 24 weeks after the end of treatment (9- month total)

Exclusion Criteria:

1. Significant cognitive impairment
2. Women who are pregnant (does not impact eligibility post study initiation)
3. Actively suicidal or homicidal
4. Active psychosis and/ or
5. Unstable medical conditions that contraindicate proposed treatment

Subject Exit criteria:

1. Increases in alcohol or drug use leading to the need for a more intensive level of care (i.e., medical detoxification, inpatient)
2. Newly developed active suicidal or homicidal ideation
3. Inability to manage psychiatric symptoms within the inclusion/exclusion criteria of the study (i.e., need for the initiation of maintenance psychotropic medications; development of psychosis). If it is determined, based on clinical criteria, that a participant needs to be started on maintenance medications for anxiety, mood or psychotic symptoms during the study, they will be discontinued from the treatment trial
4. Inability to return for therapy sessions for four consecutive weeks.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Adherence Rate | 9 months
  Adherence rate operationalized as number of weeks a participant continually receives MOUD as prescribed by primary provider for the duration of the intervention and follow-up period

SECONDARY OUTCOMES:
Relapse | 9 months
  Relapse as measured through both self-report utilizing the Timeline Follow-Back (TLFB) and Urine Drug Screen (UDS). The TLFB is a structured interview using calendar-based anchors to assess weekly drug use. UDS is a weekly urine dipstick for substance use; the urine cup has a multi-drug 12 panel test on the cup's surface, which detects several substances including opiates, and uses concentrations levels established by SAMSHA. A participant will be coded as positive for use (i.e., having relapsed) if: (a) the participant self-reported use for that week; or (b) the participant denied use, but provided a positive urine drug screen for opioids. Relapse will be ascertained in 30-day periods. At baseline, a Timeline Followback (TLFB)8 for the 30 days before admission will be obtained (with opioid use separated from other drug use) and a urine drug screen collected. For follow-up assessments, the TLFB for the previous 60 days, 3 months, 3 months post and 6 months post will be obtained.
Cravings | 9 months
  Cravings as measured by the Opioid Craving Scale (OCS), a modification of the Cocaine Craving Scale will be utilized to assess opioid craving. The OCS consists of three items rated on a visual analogue scale from 0-10: (1) How much do you currently crave opiates? (rated from not at all to extremely), (2) In the past week, please rate how strong your desire to use opiates has been when something in the environment has reminded you of opiates (rated from no desire to extremely strong), and (3) Please imagine yourself in the environment in which you previously used opiates. If you were in this environment today and if it were the time of day that you typically used opiates, what is the likelihood that you would use opiates today? (rated from not at all to I'm sure I would use opiates). The total score is calculated by averaging the three items.
Depression | 9 months
  Depression as measured by the Patient Health Questionnaire (PHQ-9), a 9-item self-report that measures depressive symptoms
Stress | 9 months
  Stress as measured by the Perceived Stress Scale (PSS), a 10-item self-report of perceived stress
Anxiety | 9 months
  Anxiety as measured by the Generalized Anxiety Disorder Scale (GAD-7), a 7-item self-report of anxiety
Quality of Life | 9 months
  Quality of life as measured by the PROMIS Physical Functioning/ Quality of Life, a 6-item self report of physical functioning and quality of life

OTHER OUTCOMES:
Cortisol Reactivity | 9 months
  Cortisol reactivity to drug cues as measured by non-invasive salivary cortisol levels. Non-invasive salivary cortisol levels will be assessed as a measure of stress reactivity to cues at baseline, post-treatment, and follow-up time points. Two samples will be acquired at each assessment session to represent resting baseline cortisol levels, stress induced cortisol levels to drug-related cues, and return to rest levels. To minimize diurnal cycle effects, assessment will take place in the afternoon when cortisol is lower, and reactivity can be detected. After 20 minutes at rest, five mL of saliva will be collected via the passive drool. Next, participants will watch a 20-minute video depicting drug cues. A second sample will then be collected to assess cortisol reactivity to drug cues. Participants will be asked to rate the extent of high, craving, and withdrawal feelings using a 10-point scale. Samples will be transported in coolers to Dr. Glenn's lab where they will be immediately

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Birmingham Veteran Affairs Medical Center, Birmingham, Alabama
  - Pathway Healthcare, LLC, Birmingham, Alabama
  - Tuscaloosa Veteran Affairs Medical Center, Tuscaloosa, Alabama
  - University of Alabama, Tuscaloosa, Alabama

IPD SHARING:
Plan to Share IPD: Undecided